CLINICAL TRIAL: NCT04583735
Title: A Phase 4, Randomized, Double-masked, Placebo-controlled, Multicenter Trial to Evaluate the Efficacy and Safety of TEPEZZA® in Treating Patients With Chronic (Inactive) Thyroid Eye Disease
Brief Title: A Study Evaluating TEPEZZA® Treatment in Patients With Chronic (Inactive) Thyroid Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZNP-TEP-403
Record Dates: First submitted 2020-10-06; First posted 2020-10-12 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Thyroid Eye Disease; Chronic (Inactive) Thyroid Eye Disease
Keywords: Proptosis
MeSH Terms: conditions — Graves Ophthalmopathy; Bronchiolitis Obliterans Syndrome; Sedentary Behavior; Exophthalmos | interventions — teprotumumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEPEZZA (Other): Participants received intravenous infusion of 10 milligrams per kilogram (mg/kg) teprotumumab at first infusion and then 20 mg/kg once every 3 weeks (Q3W) for next 7 infusions during the double masked treatment period. Proptosis non-responders who completed the double-masked treatment period had opted to receive 10 mg/kg teprotumumab at first infusion and then 20 mg/kg Q3W for next 7 infusions during open label treatment period.
  Interventions: Biological: TEPEZZA
- Placebo (Placebo Comparator): Participants received teprotumumab matching placebo by intravenous infusion, Q3W for 8 infusions during the double masked treatment period. Proptosis non-responders who completed the double-masked treatment period had opted to receive 10 mg/kg teprotumumab at first infusion and then 20 mg/kg Q3W for next 7 infusions during open label treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: TEPEZZA — Intravenous infusion
  Other Names: teprotumumab-trbw; HZN-001
  Arms: TEPEZZA
Drug: Placebo — Intravenous infusion
  Other Names: sodium chloride
  Arms: Placebo

SUMMARY:
The overall objective is to investigate the efficacy, safety and tolerability of TEPEZZA® in participants with chronic (inactive) TED (thyroid eye disease). Approximately 57 participants will be enrolled. There will be a treatment period (through Week 24) and a follow up period (where TEPEZZA will not be infused).

DETAILED DESCRIPTION:
This is a randomized, double-masked, placebo-controlled, parallel-group, multicenter trial. Participants will be screened for the trial within 4 weeks prior to Baseline (Day 1). Approximately 57 participants who meet the trial eligibility criteria will be randomized on Day 1 in a 2:1 ratio to receive 8 infusions of TEPEZZA or placebo once every 3 weeks.

All participants will enter a 24-week double-masked Treatment Period, during which trial drug will be infused on Day 1 (Baseline) and Weeks 3, 6, 9, 12, 15, 18 and 21 (with a final visit at Week 24 of the 24-week Treatment Period). At the end of the double-masked Treatment Period (Week 24), all patients will be assessed for treatment response. Non-responders may choose to receive 8 infusions of TEPEZZA in an open-label fashion q3W at Weeks 24, 27, 30, 33, 36, 39, 42 and 45.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female at least 18 years old at Screening.
3. Initial diagnosis of TED ≥2 years but <10 years prior to Screening. Clinical diagnosis of stable, chronic (inactive) TED, as determined by participant medical records indicating a Clinical Activity Score (CAS) ≤1 in both eyes for at least 1 year prior to Screening or all of the following:

   1. no progression in proptosis for at least 1 year prior to Screening
   2. if participant has history of diplopia due to TED, no progression in diplopia for at least 1 year prior to Screening
   3. no new inflammatory TED symptoms for at least 1 year prior to Screening
4. CAS ≤1 at the Screening and Baseline Visits.
5. Proptosis ≥3-mm increase from participant's Baseline (prior to diagnosis of TED), as estimated by treating physician and/or proptosis ≥3 mm above normal for race and gender.
6. Participants must be euthyroid with the participant's Baseline disease under control or have mild hypo- or hyperthyroidism (defined as free thyroxine and free triiodothyronine levels <50% above or below the normal limits) at Screening. Every effort should be made to correct the mild hypo- or hyperthyroidism promptly and to maintain the euthyroid state for the full duration of the trial.
7. Does not require immediate surgical ophthalmological intervention and is not planning corrective surgery/irradiation during the course of the trial.
8. Diabetic participants must have HbA1c ≤8.0% at Screening.
9. Participants with a history of inflammatory bowel disease, ulcerative colitis or Crohn's disease must be in clinical remission for at least 3 months, with no history of bowel surgery within 6 months prior to screening and no planned surgery during the trial. Concomitant stable therapies for inflammatory bowel disease without modifications in the 3 months prior to Screening are allowed.
10. Women of childbearing potential (including those with an onset of menopause <2 years prior to Screening, non-therapy-induced amenorrhea for <12 months prior to Screening, or not surgically sterile [absence of ovaries and/or uterus]) must have a negative serum pregnancy test at Screening and negative urine pregnancy tests at all protocol-specified time points (i.e., prior to each dose and throughout participant's participation); participants who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the trial, 1 of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started at least 1 full cycle prior to Baseline and continue for 180 days after the last dose of trial drug. Highly effective contraceptive methods (failure rate <1% per year), when used consistently and correctly, include implants, injectables, combination oral contraceptives, some intrauterine devices, sexual abstinence and vasectomized partner.
11. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.

Exclusion Criteria:

1. Decreased best-corrected visual acuity due to optic neuropathy, defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect or color defect secondary to optic nerve involvement within the last 6 months.
2. Corneal decompensation unresponsive to medical management in the study eye
3. Decrease in proptosis of ≥2 mm in the study eye between Screening and Baseline.
4. Prior orbital irradiation, orbital decompression in the study eye.
5. Prior strabismus surgery.
6. Alanine aminotransferase or aspartate aminotransferase >3 × the upper limit of normal or estimated glomerular filtration rate ≤30 mL/min/1.73 m2 at Screening.
7. Use of any steroid (IV, oral, steroid eye drops) for the treatment of TED or other conditions within 3 weeks prior to Screening. Steroids cannot be initiated during the trial. Exceptions include topical and inhaled steroids and steroids used to treat infusion reactions.
8. Any treatment with rituximab (Rituxan® or MabThera®) within 12 months prior to the first infusion of trial drug or tocilizumab (Actemra® or Roactemra®) within 6 months prior to the first infusion of trial drug. Use of any other non-steroid immunosuppressive agent within 3 months prior to the first infusion of trial drug.
9. Any previous treatment with TEPEZZA, including previous enrollment in this trial or participation in a prior teprotumumab trial.
10. Treatment with any mAb within 3 months prior to Screening.
11. Identified pre-existing ophthalmic disease that, in the judgment of the Investigator, would preclude trial participation or complicate interpretation of trial results.
12. Use of an investigational agent for any condition within 60 days or 5 half-lives, whichever is longer, prior to Screening or anticipated use during the course of the trial.
13. Malignant condition in the past 12 months (except successfully treated basal/squamous cell carcinoma of the skin or cervical cancer in situ).
14. Pregnant or lactating women.
15. Current drug or alcohol abuse or history of either within the previous 2 years, in the opinion of the Investigator or as reported by the participant.
16. Known hypersensitivity to any of the components of TEPEZZA or prior hypersensitivity reactions to mAbs.
17. Poorly controlled human immunodeficiency virus infection or untreated or positive viral load for hepatitis C or hepatitis B infections.
18. Any other condition that, in the opinion of the Investigator, would preclude inclusion in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (12):
  - The Private Practice of Raymond Douglas, Beverly Hills, California
  - Perlman Medical Offices / UCSD, La Jolla, California
  - MACRO Trials, Los Angeles, California
  - Univ of Colorado Dept of Ophthalmology, Aurora, Colorado
  - Bascom Palmer Eye Institute / Univ of Miami, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Las Vegas Endocrinology, Las Vegas, Nevada
  - Endocrinology Specialists & Thyroid Center, Greenville, South Carolina
  - Hamilton Eye Institute / U Tennessee, Memphis, Tennessee
  - Neuro-Eye Clinical Trials, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: Related Info — http://www.TEPEZZA.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Results reported are for double-masked treatment period (24 weeks) based on the primary completion date of 17 Mar 2023. Study consisted of double-masked treatment period (Week 24) and open label treatment period (Week 48).
Groups:
- Teprotumumab: Participants received intravenous infusion of 10 milligrams per kilogram (mg/kg) teprotumumab at first infusion and then 20 mg/kg once every 3 weeks (Q3W) for next 7 infusions during the double masked treatment period. Proptosis non-responders who completed the double-masked treatment period had opted to receive 10 mg/kg teprotumumab at first infusion and then 20 mg/kg Q3W for next 7 infusions during open label treatment period.
Period: Double-masked Treatment Period
Arm/Group | Teprotumumab | Placebo
Started | 42 | 20
Intent-to-treat Populaton | 42 | 20
Safety Analysis Population | 41 | 20
Completed | 39 | 19
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open-label Treatment Period
Arm/Group | Teprotumumab | Placebo
Started | 12 (All participants who completed double blind period did not enter the open label period) | 12 (All participants who completed double blind period did not enter the open label period)
Completed | 10 | 10
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants to receive study drug.
Groups:
- Teprotumumab: Participants received intravenous infusion of 10 mg/kg teprotumumab at first infusion and then 20 mg/kg Q3W for next 7 infusions during the double masked treatment period. Proptosis non-responders who completed the double-masked treatment period had opted to receive 10 mg/kg teprotumumab at first infusion and then 20 mg/kg Q3W for next 7 infusions during open label treatment period.
- Total: Total of all reporting groups
Arm/Group | Teprotumumab | Placebo | Total
Number analyzed (Participants) | 42 | 20 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (14.37) | 49.0 (16.45) | 48.7 (14.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 18 | 50
  Male | 10 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 36 | 15 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 22 | 12 | 34
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Proptosis for study eye [Mean (Standard Deviation); unit: Millimeter] | 24.60 (3.007) | 24.00 (2.824) | 24.40 (2.939)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Proptosis of Study Eye at Week 24
Description: Proptosis assessments were performed using a Hertel exophthalmometer. It measures the anterior projection of the eye from the lateral orbital rim to the cornea (proptosis).
Time Frame: Baseline, week 24
Population: ITT Population with available data at specified time point
Measure: Least Squares Mean (Standard Error); unit: Millimieter (mm)
Arm/Group | Teprotumumab | Placebo
Number analyzed (Participants) | 39 | 20
Millimieter (mm) | -2.41 (0.228) | -0.92 (0.323)
Statistical Analysis 1: Comparison: Teprotumumab vs Placebo; Test type: Superiority; p = 0.0004, MMRM — MMRM analysis with an unstructured variance-covariance matrix including change from Baseline value as dependent variable & covariates: Baseline value, treatment group, visit, visit-by-treatment & visit-by-Baseline value interactions; LSMean difference = -1.48, 95% CI 2-sided [-2.28 to -0.69], Standard Error of Mean 0.396

ADVERSE EVENTS:
Time Frame: From first dose of study drug until week 24
Description: Safety population included all participants who received at least one dose of study drug.
  AE data was reported for double-masked treatment period (24 weeks) based on the primary completion date of 17 Mar 2023.
Arm/Group | Teprotumumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/20
Other Adverse Events (participants affected / at risk) | 33/41 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teprotumumab (N=41) | Placebo (N=20)
Conductive deafness (Ear and labyrinth disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 — Participant received single dose of teprotumumab for their first dose.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teprotumumab (N=41) | Placebo (N=20)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 2 (2) | 2 (3)
Hypoacusis (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 2 (3)
Blepharospasm (Eye disorders) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 5 (8) | 1 (1)
Eye pruritus (Eye disorders) | 3 (3) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (12) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Fatigue (General disorders) | 9 (11) | 2 (3)
Feeling of body temperature change (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 2 (2)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 3 (3) | 0 (0)
Human chorionic gonadotropin increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (20) | 3 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Dysgeusia (Nervous system disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT04583735/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT04583735/SAP_001.pdf